CLINICAL TRIAL: NCT04083079
Title: Cost-Effectiveness Study of Pegylated Recombinant Human Granulocyte Colony-stimulating Factor(PEG-rhG-CSF) in Prophylactic Treatment of Neutropenia After Chemotherapy in Lymphoma
Brief Title: Cost-Effectiveness Study of PEG-rhG-CSF in Prophylactic Treatment of Neutropenia After Chemotherapy in Lymphoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director，Hematology Department, Ruijin Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEG-rhG-CSF-01
Record Dates: First submitted 2019-08-26; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Lymphoma, Non-Hodgkin; Granulocyte Colony-Stimulating Factor; Cost-Benefit Analysis
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEG-rhG-CSF cohort (Experimental): PEG-rhG-CSF primary/secondary prevention will be given 24-72 hours after each cycle for only once.
  Dosage: 6mg for weight ≥45kg，3mg for weight <45kg, subcutaneous injection
  Interventions: Drug: PEG-rhG-CSF
- rhG-CSF cohort (Experimental): rhG-CSF primary/secondary prevention will be given 24-72 hours after each cycle until absolute neutrophil count ≥2×10^9/L.
  rhG-CSF treatment will be given when there is neutropenia until absolute neutrophil count ≥2×10^9/L.
  Dosage: 5μg/kg/d, subcutaneous injection
  Interventions: Drug: rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF — Patients will be given PEG-rhG-CSF for primary/secondary prevention each cycle.
  Arms: PEG-rhG-CSF cohort
Drug: rhG-CSF — Patients will be given rhG-CSF for either primary/secondary prevention or treatment once any neutropenia each cycle.
  Arms: rhG-CSF cohort

SUMMARY:
This is a pharmacoeconomic research to explore the cost-effectiveness of PEG-rhG-CSF and rhG-CSF in prophylactic treatment of neutropenia in lymphoma patients. It should provide more scientific basis for clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* histologically confirmed de novo Non Hodgkin's lymphoma (except highly aggressive lymphoma such as lymphoblastic lymphoma and Burkitt lymphoma)
* plan to be given 6-8 cycles of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) ± Rituximab (R)
* KPS ≥70
* plan continuous PEG-rhG-CSF or rhG-CSF adiministration after at least 3 cycles of treatment for neutropenia prophylactic treatment
* absolute neutrophil count≥1.5×109/L，platelet count ≥100× 109/L，hemoglobin≥90g/L，while blood cell count≥3.0×109/L，without bleeding signs
* adquate liver and renal function as protocol discribed
* no serious cardiovascular disease as protocol discribed
* under good mental conditions and informed consented
* potential benefit for subjects based on investigators' decision

Exclusion Criteria:

* history of hematopoetic stem cell transplantationor organ transplantation
* uncontrollable infection
* allergic to study drugs or ingredients
* accepted any other investigational drug or participated another interventional study within 30 days during screening period
* other uncontrollable conditions judged by the investigator
* breast-feeding , pregnant or plan to be pregnant during study observation period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Incremental Cost-Effectiveness ratio | 1 year
  A comparison of the different strategies based on the incremental cost-effectiveness ratio (ICER), which is defined by the difference in costs between interventions, divided by the difference in their measured impact

SECONDARY OUTCOMES:
Cost-Effectiveness ratio | 1 year
  A comparison of the different strategies based on the cost-effectiveness ratio (ICER), which is defined by the difference in costs between interventions, divided by the difference in their measured impact
Sensitivity analysis | 1 year
  A sensitivity analysis is a way of examining Sensitivity to Change in results due to changes in the parameter values applied within a certain scope.
Incidence of febrile neutropenia | 1 year
  Incidence of febrile neutropenia （i.e. absolute neutrophil count<0.5×10^9/L and temperature ≥38℃）in each cycle
Duration time of febrile neutropenia | 1 year
  Duration time of febrile neutropenia （i.e. absolute neutrophil count<0.5×10^9/L and temperature ≥38℃）in each cycle
Incidence of grade 3-4 neutropenia | 1 year
  Incidence of grade 3-4 neutropenia（i.e. absolute neutrophil count<1×10^9/L）in each cycle
Duration time of grade 3-4 neutropenia | 1 year
  Duration time of grade 3-4 neutropenia（i.e. absolute neutrophil count<1×10^9/L）in each cycle
Relative dosage intensity | 1 year
  comparison between planned and actual chemotherapy dosage in each cycle
Usage rate of antibiotics | 1 year
  Usage rate of antibiotics during study period
Adverse events | 1 year
  incidence and severity of adverse events during study period

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital, Shanghai, Shanghai Municipality, China